CLINICAL TRIAL: NCT06853587
Title: Pharmacogenetic-Guided Antidepressant Prescribing in Adolescents With Anxiety and Depression
Acronym: PGx-GAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Chad Bousman, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-23-0532
Record Dates: First submitted 2025-02-20; First posted 2025-03-03 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-02

CONDITIONS: Anxiety and Depression
Keywords: depression; anxiety; adolescence; SSRI; antidepressant; pharmacogenetics
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This is a parallel arm randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, their prescribing physician, and the investigator will all be blinded to study arm. The study coordinator will be the only one unblinded to study arm allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Pharmacogenetic (PGx)-Guided (Experimental): Participants and their physician will receive a one-time prescribing report after completing baseline for selective serotonin reuptake inhibitors with dosing information based on CYP2B6, CYP2C19, and CYP2D6 genotype data, and clinical practice guidelines for fluoxetine as there are no pharmacogenetic guidelines for this medication.
  Interventions: Other: Pharmacogenetic-guided dosing
- Current Prescribing Guidelines/Recommendations (Active Comparator): Participants and their physician will receive a one-time prescribing report after completing baseline for selective serotonin reuptake inhibitors based on current prescribing guidelines/recommendations.
  Interventions: Other: Current prescribing guidelines/recommendations

INTERVENTIONS:
Other: Pharmacogenetic-guided dosing — SSRI dosing based on Clinical Pharmacogenetics Implementation Consortium's SSRI dosing guidelines.
  Arms: Experimental: Pharmacogenetic (PGx)-Guided
Other: Current prescribing guidelines/recommendations — SSRI dosing based on current prescribing guidelines/recommendations
  Arms: Current Prescribing Guidelines/Recommendations

SUMMARY:
This is a parallel arm randomized (1:1) controlled trial. Adolescents aged 12-17 years (n=452) who are starting or changing a selective serotonin reuptake inhibitor (SSRI) for depression and/or anxiety will be randomly allocated to receive 12-weeks of pharmacogenetic-guided antidepressant therapy (experimental intervention) or current prescribing guidelines/recommendations guided therapy (control intervention).

DETAILED DESCRIPTION:
Goal: To test the efficacy of pharmacogenetic-guided antidepressant prescribing for adolescents with depression.

Background: For an adolescent with depression and anxiety, antidepressant medication is prescribed, often in combination with psychotherapy. The class of antidepressants recommended for use is selective serotonin reuptake inhibitors (SSRIs) with fluoxetine recommended as the first-line medication, and four other SSRIs recommended for consideration (sertraline, citalopram, escitalopram, fluvoxamine) if the adolescent does not respond or tolerate fluoxetine. For most adolescents, medication prescribing, and monitoring will be managed by a primary care physician or community pediatrician rather than by a mental health care provider, and guidelines exist to support this management. However, current prescribing guidelines/recommendations do not account for SSRI metabolism phenotypes that could change whether the SSRI selected is efficacious or tolerated. Our team of researchers, clinician scientists, patient partners, and primary care providers has designed a trial to test the impact of accounting for metabolism phenotypes, through pharmacogenetic-guided antidepressant prescribing, on adolescent outcomes, experiences, and health care utilization.

Principal Question: Compared to current prescribing guideline/recommendation informed prescribing, does pharmacogenetic-guided prescribing for adolescents with depression and/or anxiety have superior efficacy following 12-weeks of therapy with a SSRI?

The Trial: This is a parallel arm randomized controlled trial. Adolescents aged 12-17 years (n=452) who are starting or changing a SSRI for depression and/or anxiety will be randomly allocated to receive pharmacogenetic-guided antidepressant therapy (experimental intervention) or current prescribing guideline/recommendation guided prescribing (control intervention). Participants and prescribing physicians will be blinded to which intervention was received. The primary outcome is depressive symptom remission at 12 weeks measured using the Quick Inventory of Depressive Symptomatology - Adolescent (17-item) (QIDS-A17) and anxiety symptom remission at 12 weeks measures using the Screen for Child Anxiety Related Disorders (SCARED). Secondary outcomes include side effects, role functioning, medication adherence, and health-related quality of life measured 4-, 8-, and 12-weeks after intervention initiation as well as cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-17
* Depression and/or anxiety as the primary concern, confirmed by the treating physician
* Intention to start a new SSRI
* English fluency

Exclusion Criteria:

* Co-occurring obsessive compulsive disorder, psychosis, bipolar disorder, eating disorder, autism spectrum disorder, fetal alcohol spectrum disorder, or intellectual disability
* History of non-response to 3 or more SSRI medications as confirmed by the treating physician
* Brain stimulation-based therapy initiated within 8 weeks of referral, or plans to initiate/change brain stimulation during study participation
* History of liver or hematopoietic cell transplant
* History of CYP2B6, CYP2C19, or CYP2D6 testing

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 452 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with depression remission | Baseline to 12 weeks
  Quick Inventory of Depressive Symptomatology - Adolescent - 17-item (QIDS-A17) total score < 6. Scores range from 0-27, with higher scores indicative of more severe depression.
Number of participants with anxiety remission | Baseline to 12 weeks
  Screen for Child Anxiety Related Disorders (SCARED) total score < 25. Scores range from 0-82, with higher scores indicative of more severe anxiety.

SECONDARY OUTCOMES:
Number of participants with side effects and adverse drug reactions | Baseline to 12 weeks
  Frequency, Intensity, Burden of Side Effects Rating (FIBSER) scale. Total scores range from 0-6 (3 items); cut-points are used to indicate moderate (score of 3) or severe (score of 5) adverse drug reaction/side effect interference with activities.
Percent change in role functioning | Baseline to 12 weeks
  WHO Disability Assessment Schedule. Scores range from 0 to 48, with higher scores indicative of worse role functioning.
Percent change in depressive symptom severity | Baseline to 12 weeks
  Quick Inventory of Depressive Symptomatology - Adolescent - 17-item (QIDS-A17). Scores range from 0-27, with higher scores indicative of more severe depression.
Percent change in anxiety symptom severity | Baseline to 12 weeks
  Screen for Child Anxiety Related Disorders (SCARED) total score < 25. Scores range from 0-82, with higher scores indicative of more severe anxiety.
Percent change in clinician assessment of depressive and anxiety symptom severity | Baseline to 12 weeks
  Change in Clinical Global Impression Severity (CGI-S) scale. Scores range from 0-7, with higher scores indicative of more severe illness.
Change in self-report health care resource use | Baseline to 12 weeks
  Resource use questionnaire that captures number of visits and out-of-pocket costs for various mental health services.
Change in healthcare utilization - physician visits | Baseline to 12 weeks
  Administrative data will be obtained on change in number of physician visits.
Change in health care utilization - emergency department visits | Baseline to 12 weeks
  Administrative data will be obtained on change in number of emergency department visits.
Change in health care utilization - hospitalizations | Baseline to 12 weeks
  Administrative data will be obtained on change in number of hospitalizations.
Change in prescribed medication dose | Baseline to 12 weeks
  Administrative data will be obtained on changes to prescribed medication doses.
Change in prescribed agent | Baseline to 12 weeks
  Administrative data will be obtained on changes of agent for prescribed medications.
Change in prescribed medication duration | Baseline to 12 weeks
  Administrative data will be obtained on duration of use of prescribed medications.
Change in health-related quality of life | Baseline to 12 weeks
  EuroQoL 5 Dimension - Youth (EQ-5D-Y). Five descriptive items code level of perceived problems in health states and a visual analog scale has a score from 0-100, with higher scores indicative of better health.
Change in medication adherence | 4 to 12 weeks
  Medication Adherence Report Scale (MARS-5) scores. Scores range from 5-25 with higher scores indicative of better medication adherence.
Change in behavioral activation | Baseline to 12 weeks
  Emergence of activation based on Treatment-Emergent Activation and Suicidality Assessment Profile. Total scores range from 0-114 (38 items) with higher scores indicating greater behavioral activation.

OTHER OUTCOMES:
Minimally clinically important differences | 12 weeks
  Participant-reported, Global Rating of Change Scale (GRCS) (11-point Likert scale ranging from +5 to -5) to indicate the degree to which symptoms and role functioning changed for the better, for the worse, or no change was experienced.
Intervention fidelity | 12 weeks
  Physician-reported, two questions on use of recommendations in the dosing report.
Blinding fidelity | 12 weeks
  Physician-reported, 1-item survey about the perceived allocation of each of their participating patients; response options are 'PGx-guided prescribing', 'don't know' or 'current prescribing guidelines/recommendations'

CONTACTS AND LOCATIONS:
Overall Officials: Chad Bousman, PhD, Principal Investigator — University of Calgary; Amanda Newton, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized, individual participant PGx-GAP data will be shared using a controlled-access model. Under this model, the data will be released to a researcher if access criteria are met.
  All requests for data sharing should be made to the Co-Principal Investigators who will be responsible for reviewing and granting requests. Requestors should provide a research proposal for review. In the event that a data sharing request is declined, reasons will be provided to the requestor. If the data sharing request is granted, a data-sharing agreement will be initiated by the Co-Principal Investigators alongside the University of Calgary (lead institution). This agreement will include information on the individual data to be shared; if other documents will be available (e.g., statistical codes, data dictionary), when the data will be available and for how long, and how data access will be provided (e.g., file transfer).
Access Criteria: 1. The requestor is affiliated with an academic institution as an independent investigator or trainee of an independent investigator;
  2. The proposed research question(s) and hypothesis(es) are specific, measurable, and achievable;
  3. The proposed research project will be governed/overseen by a local legal/regulatory body;
  4. The proposed research project poses no risk of invasion of privacy or breaches of confidentiality for trial participants;
  5. A member of the proposed research team has sufficient statistical skills to carry out the proposed analytic plan;
  6. The requestor has sufficient financial and/or human resources to see the proposed research project to completion;
  7. The proposed research question(s) and hypothesis(es) do not conflict with active or planned studies of the Co-Principal Investigators.